CLINICAL TRIAL: NCT06702358
Title: Potential Therapeutic Implications of Laser Acupoints on Visceral Fat and Hormonal Changes in Post-menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Nawal Reda Rashad Mohamed, DEPARTEMENT OF PHYSICAL THYRAPY FOR WOMAN'S HEALTH, Kafrelsheikh University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-92
Record Dates: First submitted 2024-11-07; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Post-menopausal Women; Visceral Fat

STUDY DESIGN:
Intervention Model Description: Laser pointer instruments Product Details Infrared laser diode made in Italy, it must be perpendicular with direct contact to each point.
  Each point will stimulate bilaterally by a laser beam of the following parameters wave length 904 nm; strength, 24 mW; energy, 0.1 J; stimulation time, 30 s/point; and two sessions per week for 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infrared laser diode (Other): Laser pointer instruments Product Details Infrared laser diode made in Italy, it must be perpendicular with direct contact to each point.
  Each point will stimulate bilaterally by a laser beam of the following parameters wave length 904 nm; strength, 24 mW; energy, 0.1 J; stimulation time, 30 s/point
  Interventions: Other: Potential Therapeutic Implications of laser Acupoints on Visceral Fat and Hormonal Changes in Post-menopausal Women

INTERVENTIONS:
Other: Potential Therapeutic Implications of laser Acupoints on Visceral Fat and Hormonal Changes in Post-menopausal Women — Application of laser acupuncture ( E M E ) on 10 acupuncture procedure for each woman which will be detected by therapist according to Acupuncture points Will stimulate St 25 (Tianshu), St 36 (Zusanli), Liv 3 (Taichong); P 6 (Neiguan), H 7 (Shenmen) for the psychical aspect of the therapy and Auriculothera- py: 55 (Shenmen) and 87 (Stomach) Each point stimulating will be Stimulation time, 30 s/point

SUMMARY:
Potential Therapeutic Implications of laser Acupoints on Visceral Fat and Hormonal Changes in Post-menopausal Women

DETAILED DESCRIPTION:
All the patients fitted the inclusion criteria, will be given explanation of the treatment protocol in their understandable language.

Treatment procedures. Group (A): will receive laser acupuncture in addition to traditional treatment (low calorie-diet and physical activity) Group (B): will receive traditional treatment only

Laser acupuncture technique:

Application of laser acupuncture on 10 acupuncture procedure for each woman which will be detected by therapist according to Acupuncture points Will stimulate St 25 (Tianshu), St 36 (Zusanli), Liv 3 (Taichong); P 6 (Neiguan), H 7 (Shenmen) for the psychical aspect of the therapy and Auriculothera- py: 55 (Shenmen) and 87 (Stomach) Each point stimulating will be Stimulation time, 30 s/point two sessions per week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women
* Woman with visceral obesity
* with age ranges from 50-65years
* Body mass index (BMI) more than 30 kg/m2
* WHR more than 0.8

Exclusion Criteria:

* Endometrial cancer

  * Insulin resistance
  * Or metabolic disorders
* Diabetes
* Hypertensive •NOT receiving any medication of obesity

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Post-menopausal Women
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Potential Therapeutic Implications of laser Acupoints on Visceral Fat and Hormonal Changes in Post-menopausal Women | for 8 weeks
  measured in both group before and after treatment. To get in touch with the hunger and satiety cues,BMI ,WHR and serum insulin level.
Body Mass Index (BMI) | for 8 weeks
  The weight in kg

CONTACTS AND LOCATIONS:
Locations (1):
- Nawal Reda Rashad Mohamed, Cairo, US, Egypt